CLINICAL TRIAL: NCT01752062
Title: Observational Study of Conception/Pregnancy in Adult Patients With Chronic Myeloid Leukemia (CML) Treated With Tyrosine Kinase Inhibitors
Brief Title: Observational Study of Conception/Pregnancy in Adult Patients With CML Treated With Tyrosine Kinase Inhibitors
Acronym: CML1012
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: CML1012
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Chronic Myeloid Leukemia; Pregnancy
Keywords: Chronic Myeloid Leukemia; CML; Pregnancy
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to acquire more information about what we are doing during pregnancy in CML patients, in order to possibly establish in the future a consensus on the management of patients receiving TKIs who wants to father a child or become/are pregnant.

DETAILED DESCRIPTION:
The management of patients with chronic myeloid leukemia (CML) during pregnancy is a matter of continued debate. The introduction of the TKIs in clinical practice has dramatically changed the prognosis of CML. Patients diagnosed in chronic phase can reasonably expect many years of excellent disease control and good quality of life. Thus, the need to address issues related to fertility and pregnancy have arisen. Physicians are frequently being asked for advice regarding the need for, and or the appropriateness of, stopping treatment in order to conceive. The management of fertility begins at diagnosis. This means that immediate and future treatments should be considered at the very beginning. Therefore, the maintenance of fertility should be taken into account since diagnosis. Imatinib is not genotoxic but might lead to a decrease in sperm counts. Nevertheless, Imatinib is teratogenic in rats when given during organogenesis at doses higher than 100 mg/kg, approximately equivalent to 800 mg/day in men. Until now, approximately 60 pregnancies were reported in partners of men on Imatinib. No suggestions of any problems in conception, pregnancy, delivery or any increase in congenital abnormalities were reported. Regarding women, 204 patients were exposed to Imatinib, and 180 were reported in literature (76, 77). Of 180 women exposed to imatinib during pregnancy, outcome data are available for 125 (69%). Of those with known outcomes, 50% delivered normal infants and 28% underwent elective terminations, 3 following the identification of abnormalities. There were a total of 12 infants in whom abnormalities were identified, 3 of which had strikingly similar complex malformations that are clearly a cause for concern. It appears that although most pregnancies exposed to imatinib are likely to have a successful outcome, there remains a risk that exposure may result in serious fetal malformations. Although numbers are small there has been a disturbing cluster of rare congenital malformations such that imatinib cannot be safely recommended, particularly during the period of organogenesis. Last but not least, it has recently been reported a poor outcome after reintroduction of Imatinib in patients who interrupt therapy for pregnancy without having achieved an optimal response (78), introducing another variable in the management of women pregnant while receiving Imatinib. Only few data are available about the use of second generation TKIs, Nilotinib and Dasatinib, during pregnancy. Dasatinib is not mutagenic in rats (in vitro and in vivo tests), but is clastogenic in CHO cells. It does not seem to have such effect on fertility of male and female rats. However, it gives skeletal alterations in rats and rabbits and has embryolethality in rats if administered during pregnancies. Eleven pregnancies were reported while in dasatinib: 5 patients delivered normal infants, while 3 elective termination and 2 spontaneous abortion were reported. On the other hand, 9 male patient conceived during dasatinib: 8 normal infants were delivered, and 1 case was ongoing at the time of the report. Nilotinib is not mutagenic in rats. It does not have any effect on fertility in male and female rats. When administered during pregnancy, there is no evidence of teratogenicity but it is embryo and foetotoxic in the rat and in the rabbit. Only sporadic cases of patients who had been pregnant/had conceived during Nilotinib have been reported, and no speculation should be made from these data. In summary, there are virtually no data regarding II generation TKIs, that must be discontinued by women wishing to become pregnant. Several questions still remains unanswered regarding the management of patients receiving TKIs who want to conceive, or who have been exposed to TKI during pregnancy/conception.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Ph+/BCR-ABL+ CML in any phase of disease;
* Conception/pregnancy while diagnosed with CML
* Treatment with TKIs (before or after pregnancy);
* Signed written informed consent according to ICH/EU/GCP and national local laws.

Exclusion Criteria:

* Patient < 18 years
* Patients that suffer from any condition or illness that could prevent the patient to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (>18 years old) patients with a diagnosis of chronic myeloid leukemia (CML) who had been pregnant / had conceived while diagnosed with CML and treated with TKIs.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2013-05-02 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of normal birth, elective termination and spontaneous abortion | At 3 years from study entry
  Pregnancy outcome: it will be calculated in terms of normal birth, elective termination, spontaneous abortion
Number of patients with major molecular remission loss | At 3 years from study entry
  Cumulative Incidence of MMR loss: it will be calculated from the date of achievement of MMR using the cumulative incidence method, where death will be considered as competing risk. Patients still alive, in first MMR, will be censored at the moment of last follow-up.
Number of patients with disease progression | At 3 years from study entry.
  Cumulative Incidence of Disease Progression: it will be calculated from the date of diagnosis using the cumulative incidence method, where death without signs of disease progression will be considered as competing risk. Patients still alive, without a date of progression, will be censored at the moment of last follow-up.
Number of patients with CCgR loss | At 3 years from study entry
  Cumulative Incidence of CCgRloss: it will be calculated from the date of achievement of CCgR using the cumulative incidence method, where death in CCgR will be considered as competing risk. Patients still alive, in first CCgR, will be censored at the moment of last follow-up.

SECONDARY OUTCOMES:
Number of male and female patients conceiving during treatment | At 3 years from study entry
  Proportion of male and female patients conceiving during the treatment with TKI
Number of spontaneous abortion | At 3 years from study entry
  Proportion of spontaneous abortion
Number of of foetal abnormalities | At 3 years from study entry
  Proportion of foetal abnormalities: it will be calculated with respect to the study population and with respect to normal population.
Number of patients surviving | At 3 years from study entry
  Overall Survival (OS): it will be calculated from the date of CML diagnosis until date of death (whatever the cause). Patients still alive will be censored at the moment of last follow-up.
Number of patients alive with no disease progression | At 3 years from study entry
  Progression Free Survival (PFS): it will be calculated from the date of CML diagnosis until the date of first progression to A-B phase or until death (whatever the cause), whichever occurs first. Patients still alive, without a date of progression, will be censored at the moment of last follow-up.
Number of patients with molecular response. | At 3 years from study entry
  Duration of CCgR/ Molecular response (MR): it will be calculated from the date of achievement of CCgR, MR until first date of CCgR loss or until death (whatever the cause), whichever occurs first. Patients still alive, in first CCgR/MR, will be censored at the moment of last follow-up.
Number of patients with major molecular remission | At 3 years from study entry
  Evaluation of Major Molecular Remission (MMR)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Abruzzese, Principal Investigator — Hematology, S. Eugenio Hospital, Rome
Locations (52):
- Italy (52):
  - Unità Operativa di Oncologia - Presidio Ospedaliero N. Giannetasio - Azienda ASL 3 Rossano (CS), Rossano, Cosenza
  - Azienda Ospedaliera - Nuovo Ospedale "Torrette", Ancona
  - S.G. Moscati Hospital, Avellino
  - UO Ematologia con trapianto-Università degli Studi di Bari Aldo Moro, Bari
  - Divisione di Ematologia - Ospedali Riuniti Bergamo, Bergamo
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - Spedali Civili - Azienda Ospedaliera - U.O. Ematologia, Brescia
  - Divisione di Ematologia Ospedale A. Perrino, Brindisi
  - ASL N.8 - Ospedale "A. Businco" - Struttura Complessa di Ematologia e CTMO, Cagliari
  - Unità di Onco-Ematologia - Azienda Ospedaliera - Garibaldi, Catania
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Sezione di Ematologia e Fisiopatologia delle Emostasi - Azienda Ospedaliera - Arcispedale S. Anna, Ferrara
  - Policlinico di Careggi, Università Degli Studi Firenze, Florence
  - Clinica Ematologica - DiMI - Università degli Studi di Genova, Genova
  - Azienda Ospedaliera Universitaria - Policlinico G. Martino Dipartimento di Medicina Interna - U.O. Messina, Messina
  - Ospedale Niguarda "Ca Granda", Milan
  - UO Centro Trapianti di Midollo - IRCCS Ospedale Maggiore Policlinico, Milan
  - N. Osp. divisione di Ematologia "S.Gerardo dei Tintori", Monza
  - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli" Napoli, Napoli
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - Ospedale San Gennaro - ASL Napoli 1, Napoli
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Dip. di Scienze Cliniche e Biologiche - Ospedale S. Luigi Gonzaga-Medicina Interna 2 Prof. Giuseppe Saglio, Orbassano
  - Divisione di Ematologia con trapianto di midollo - A.U. Policlinico "Paolo Giaccone", Palermo
  - Ospedale La Maddalena - Palermo, Palermo
  - Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - Div. di Ematologia IRCCS Policlinico S. Matteo, Pavia
  - Div. di Ematologia di Muraglia - CTMO Ospedale San Salvatore, Pesaro
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Unità Operativa Ematologia e Centro Trapianti - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale di Piacenza, Piacenza
  - Università di Pisa - Azienda Ospedaliera Pisana - Dipartimento di Oncologia, dei Trapianti e delle nuove Tecnologie in Medicina - Divisione di Ematologia, Pisa
  - Ematologia - Ospedale San Carlo, Potenza
  - Ospedale S. M. delle Croci, Ravenna
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Az. Ospedaliera "Sant' Andrea"-Università la Sapienza Seconda Facoltà di Medicina e Chirurgia, Roma
  - Padiglione Cesalpino - I piano - Divisione di Ematologia - Ospedale S. Camillo, Roma
  - S.C. di Ematologia e Trapianti - I.F.O. Istituto Nazionale Tumori Regina Elena- I.F.O. Istituto Nazionale Tumori Regina Elena Roma, Roma
  - U.O.C. Ematologia - Ospedale S.Eugenio, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - UOC Pronto Soccorso e Accettazione Ematologica - Dipartimento Biotecnologie Cellulari ed Ematologia - Università degli Studi di Roma "Sapienza", Roma
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Ematologia - Dipartimento di Medicina Clinica e Sperimentale, Sassari
  - U.O.C. Ematologia e Trapianti - A.O. Senese - Policlinico " Le Scotte", Siena
  - U.O.C. di Ematolgia - A.O. " SS Annunziata" - P.O. S.G. Moscati, Taranto
  - Azienda ospedaliera S. Maria di Terni, Terni
  - SCDO Ematologia 2 AOU S. Giovanni Battista, Torino
  - Sezione di Ematologia - Med.II Div. Presidio Ospedaliero S. Chiara di Trento, Trento
  - Azienda U.L.S.S.9 - U.O. di Ematologia, Treviso
  - Policlinico Universitario - Clinica Ematologia, Udine
  - Università degli Studi di Verona - A. O. - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona
  - ULSS N.6 Osp. S. Bortolo, Vicenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GIMEMA Foundation — http://www.gimema.it